CLINICAL TRIAL: NCT03610763
Title: Harnessing Neuroplasticity to Enhance Functional Recovery in Allogeneic Hand Transplant and Heterotopic Hand Replant Recipients
Brief Title: Harnessing Neuroplasticity to Enhance Functional Recovery During Chronic Recovery From Upper Extremity Nerve Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Washington University School of Medicine (Other); Christine M. Kleinert Institute for Hand and Microsurgery (Other)
Responsible Party: Principal Investigator, Scott H Frey, PhD, Miller Family Professor of Cognitive Neuroscience, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008784; CDMRP-MR141043 (Other Grant/Funding Number: Army Medical Research & Materiel Command)
Record Dates: First submitted 2018-06-23; First posted 2018-08-01 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Hand Transplantation; Peripheral Nerve Injuries; Neurologic Rehabilitation
Keywords: Rehabilitation Neuroscience; Transcranial Direct Current Stimulation; Rehabilitation Therapy; Neuroplasticity; Transplantation; Hand Therapy; Constraint Induced Movement Therapy; Peripheral Nerve Injuries; tDCS; CIMT
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Transplantation/Replantation Patients (Active Comparator): Can plateaued hand function in hand transplantation patients/hand replantation patients in the chronic stage of recovery be facilitated by use of bi-hemispheric transcranial direct current stimulation (tDCS) combined with modified Constraint Induced Movement Therapy (CIMT)?
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Modified Constraint Induced Movement Therapy
- Nerve Injury Patients active (Active Comparator): Can plateaued hand function in peripheral nervous system injuries in the chronic stage of recovery be facilitated by use of bi-hemispheric transcranial direct current stimulation (tDCS) combined with modified Constraint Induced Movement Therapy (CIMT)?
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Modified Constraint Induced Movement Therapy
- Actigraphy Testing (No Intervention): We will acquire a set of actigraphy data from a group of hand transplant/replant patients and unilateral, adult amputees in order to evaluate typical patterns of limb use prior to hand transplantation and to investigate prosthesis utilization.

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial direct current stimulation (tDCS) is a portable neurostimulation method that modulates cortical excitability. The technique involves placing two saline-soaked electrodes (anode and cathode) on the scalp and passing a small direct current (1.5 milliamps; mA) between them. Cortex underlying the anode is more easily excited due to lowered thresholds for depolarization of glutamatergic neurons, while thresholds are increased in neurons beneath the cathode, making them less excitable. Sham stimulation is easily implemented, and the technique can be effectively double-blinded.
  Other Names: tDCS
  Arms: Nerve Injury Patients active; Transplantation/Replantation Patients
Behavioral: Modified Constraint Induced Movement Therapy — In CIMT, patients are required to wear a mitt that restricts use of the unaffected limb while they practice structured tasks and also engage in activities of daily living.
  Other Names: CIMT
  Arms: Nerve Injury Patients active; Transplantation/Replantation Patients

SUMMARY:
This study adopts a strategy that has arisen from basic neuroscience research on facilitating adaptive brain plasticity and applies this to rehabilitation to improve functional recovery in peripheral nervous system injuries (including hand transplantation, hand replantation, and surgically repaired upper extremity nerve injuries). The technique involves combining behavioral training with transcranial direct current stimulation (tDCS)-a non-invasive form of brain stimulation capable of facilitating adaptive changes in brain organization.

DETAILED DESCRIPTION:
This study will implement and evaluate an innovative program of post hand transplant rehabilitation; one that harnesses recent discoveries in neuroscience to facilitate long-term, experience-dependent adaptations within the brain's sensory and motor systems. The current approach to rehabilitation of function in allogeneic hand transplant recipients is largely the same as standard-of-care following hand replantation (re-attachment) and peripheral nerve repairs. This involves an eclectic combination of traditional therapies. In seeking to improve on this approach, there is potentially much to be gained by considering evidence that limb amputation not only impacts the peripheral nervous system but also the brain, and tailoring interventions accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Individuals whom have received a unilateral allogeneic transplantation proximal to the wrist and are at the chronic stage of recovery (approx. 12 - 18 months following surgery, when Tinel's sign reaches the distal fingertips).
* Individuals whom have undergone a complete amputation the hand between the wrist and elbow followed by successful re-attachment and are at the chronic stage of recovery (approx. 12 - 18 months following surgery, when Tinel's sign reaches the distal fingertips).
* Individuals whom have undergone repairs of the median, ulnar, or other related or nearby nerve(s) following complex volar forearm lacerations or other injuries between the distal wrist crease and the flexor musculotendinous junctions. Individuals must be at the chronic stage of recovery (approx. 12 - 18 months following surgery, when Tinel's sign reaches the distal fingertips).

Exclusion Criteria:

* Individuals with significant/severe brain trauma
* Serious psychiatric conditions
* Chronic or severe neurological conditions.
* Current pregnancy
* History of seizures or unexplained loss of consciousness
* Metallic implants above the chest
* Certain implanted medical devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Dellon Modified Moberg Pick-Up Test performance at two weeks. | Baseline, immediately after end of intervention (+/- 3 days).
  This functional test measures quality of sensibility of the hand. This outcome measure will investigate any change in participant performance between pre- and post-intervention sessions of the Dellon Modified Moberg Pick-Up Test.

SECONDARY OUTCOMES:
Change from Baseline Action Research Arm Test (ARAT) performance at two weeks. | Baseline, immediately after end of intervention (+/- 3 days).
  The Action Research Arm Test (ARAT) measures limb function by having participants pick up various objects of different sizes, different weights, and different shapes (e.g., a glass of water, a cricket ball). This secondary outcome measure will investigate any change in participant performance between pre- and post-intervention sessions of the ARAT.
Change from baseline upper limb movement as measured by actigraphy-derived variables during everyday life at periodic intervals after intervention. | Baseline, post intervention at week 1, post intervention at 1 month, post intervention at 3 months, post intervention at 6 months.
  This secondary outcome measure will employ actigraphy on participants to measure limb movement in everyday life before and after the intervention. Participants will wear wrist-watch like devices that contain accelerometers on each upper extremity in 24-72 hour sessions. Two primary variables will quantify upper limb activity from accelerometer data: the Bilateral Magnitude and the Magnitude Ratio. The Bilateral Magnitude quantifies the intensity of activity across both limbs, whereas the Magnitude Ratio quantifies the contribution of each limb to activity.
  This outcome measure will investigate the change in the Bilateral Magnitude and Magnitude Ratio between a baseline pre-intervention test and post-intervention actigraphy sessions performed within one week of completion of the intervention, at 1 month post-intervention, 3-months post intervention, and 6-months post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Scott H Frey, Ph.D., Ed.M., Principal Investigator — University of Missouri-Columbia
Locations (3):
- United States (3):
  - Christine Kleinert Institute for Hand & Microsurgery, Louisville, Kentucky
  - University of Missouri, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No